CLINICAL TRIAL: NCT03099421
Title: Prostatic Artery Embolization for Benign Prostatic Obstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Brian Malling, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-17000714-1
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Hyperplasia Prostatic; Lower Urinary Tract Symptoms; Prostatic Diseases; Urological Manifestations
Keywords: Benign prostatic obstruction; benign prostatic enlargement; benign prostatic hyperplasia; prostatic artery embolization; Quality of Life; IPSS; DAN-PSS; Complications
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms; Prostatic Diseases; Urological Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostatic Artery Embolization (Experimental): Embolization of the prostatic arteries to induce necrosis and a reduction of the prostate volume.
  Interventions: Procedure: Prostatic Artery Embolization

INTERVENTIONS:
Procedure: Prostatic Artery Embolization — The procedure is performed with the patient under local anaesthetic and if necessary sedation. We will be using a percutaneous transfemoral approach, super-selective catheterisation of small prostatic arteries is carried out using microcatheters. Embolisation will be done using microspherical embolic material.

SUMMARY:
The aim of this study is to investigate the safety and efficacy of prostatic artery embolization (PAE) for patients who refuse or are not eligible for surgery with moderate-severe lower urinary tract symptoms or indwelling catheter secondary to benign prostate obstruction due to benign prostatic hyperplasia.

DETAILED DESCRIPTION:
This is a prospective study investigating the safety and efficacy of PAE for patients who refuse or are not eligible for surgery and who suffers from moderate-severe lower urinary tract symptoms or indwelling catheter secondary to benign prostatic obstruction due to benign prostatic hyperplasia. It may form the grounding for further research in the shape of a larger randomised clinical trial.

Our hypothesis is that PAE will eliminate the need for indwelling catheter and improve IPSS 6 months post-procedure.

1, and 6 months follow-up.

Main outcome Ability to void after removal of indwelling catheter

Secondary outcomes International Prostate Symptom Score (IPSS) Quality of Life (QoL) International Index of Erectile Function (IIEF) Prostate volume Peak void flow (Qmax) Post-void residual (PVR) Classify complications according to Society of Interventional Radiology (SIR) guidelines for reporting Prostate-specific antigen (PSA)

ELIGIBILITY:
Inclusion Criteria:

* Indwelling catheter secondary to benign prostatic hyperplasia (BPH) or
* Moderate-severe Obstructive LUTS secondary to BPH refractory to medical treatment
* Unsuitable for TURP or refuse surgery

Exclusion Criteria:

* Bladder dysfunction(and known neurological conditions affecting bladder function)
* Urethral strictures
* Bladder neck contracture
* Known sphincter anomalies
* Big bladder diverticulum or stones
* Kidney insufficiency (eGFR < 45)
* Coagulation disturbances
* Severe atheromatous or tortuosity of arteries
* Allergy to contrast medium
* Unable to undergo MR imaging
* Urological malignancy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Ability to void spontaneously | 6 months
  Patient demonstrate the ability to void spontanously after the removal of the indwelling catheter at 6 months

SECONDARY OUTCOMES:
IPSS | 1, 6 months
  International Prostate Symptom Score from 0-35, 35 is most severe symptoms
QoL | 1, 6 months
  Quality of Life scored from 0-6, 6 is worst
IIEF | 1, 6 months
  International Index of Erectile Function scored from 0-25, where higher scores represents better erectile function
PV | 1, 6 months
  Prostate Volume measured by MRI
PVR | 1, 6 months
  Post-void residual
Qmax | 1, 6 months
  Peak void flow
PSA | 1, 6 months
  Prostate-specific antigen

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lönn, Professor, Study Chair — Radiologisk Klinik, Rigshospitalet
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No